CLINICAL TRIAL: NCT05625269
Title: The Effect of Education and Follow-up Program in Patients Undergoing Transcatheter Aortic Valve Implantation
Brief Title: The Effect of Education and Follow-up Program in Patients Undergoing TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Arzu AKBABA, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/26-11
Record Dates: First submitted 2022-11-07; First posted 2022-11-22 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Aortic Stenosis; Nursing Caries
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education and follow-up group (Experimental): Patients in the intervention group will be given training on the procedure and home care process on the first day of hospitalization and the day before discharge. Afterwards, patients will be followed up by phone at intervals of two weeks. The purpose of telephone monitoring is to question adherence to treatment, to identify and change barriers, to apply counseling and to control symptoms.
  Interventions: Other: Education
- Control group (No Intervention): The control group will be given the standard care applied in the clinic, and the patients of this group will be given training after the research is completed.

INTERVENTIONS:
Other: Education — The first session of the individual training will be held for the patients in the intervention group on the first day of the service hospitalization, covering the issues related to the procedure and the hospital process. Afterwards, the second session of individual education will be held the day before discharge on issues related to the patient's home care, such as treatment site care, nutrition, exercise, medication and symptom management. In addition to the patients, their families will also participate in the training sessions. The training will be given face-to-face in a quiet environment to increase intelligibility in patients' rooms. The patients will be given a booklet and magnet prepared by the researcher in addition to the oral explanation.
  Arms: Education and follow-up group

SUMMARY:
Aortic stenosis is a progressive disease that affects approximately 3% of adults aged 75 and over. If left untreated, the mortality rate of aortic stenosis, which becomes symptomatic in a short time, is 50% in the first year, while this rate rises to 90% within 5 years.

Surgical treatment of aortic stenosis has been proven to reduce symptoms and increase survival. Although surgical treatment is considered the gold standard, 30% of elderly patients cannot undergo surgery due to left ventricular dysfunction and comorbidities. The search for new methods with a low-risk rate and a more comfortable post-procedure process has begun. For this purpose, Cribier et al. Transcatheter aortic valve implantation (TAVI) was developed in 2002 as an important alternative to surgical aortic valve placement. The TAVI method; is the procedure of inserting a bioprosthetic aortic valve into the heart using the catheter method without open heart surgery.

Although transcatheter aortic valve implantation is more tolerable than surgery, it has certain complications. According to the Valve Academic Research Consortium (VARC-3), common post-procedural complications are; stroke, myocardial infarction, bleeding, major vascular complications, and acute kidney injury. Nursing-specific care problems are stated as bleeding, infection, pain, decrease in cardiac output, and sleep problems. Many factors, such as the high risk of patients undergoing TAVI, the complexity of the procedure, and the complications that may develop after the procedure, require that the nursing care to be applied be specific and individualized to the TAVI procedure. It is very important to understand the experiences of the patients to effectively carry out this special care to be applied before and after TAVI. It is known that being aware of the experiences and needs will contribute positively to the care and treatment of future patients. Instens et al. stated that experiences can be reached by examining perspectives in depth rather than clinical studies or records. In this regard, Baumbusch et al. in their qualitative design study; It has been revealed that TAVI patients cannot manage their care after the procedure because of their age and comorbidities, there is a difference between their expectations and reality, and they need support in terms of information. In another study, the post-TAVI process was defined as a balance between the struggle for life and hope, and the importance of the support of health professionals during the process was emphasized. For these reasons, TAVI patients need nursing care support and information in terms of post-procedure disease management. The most important component of successful disease management is to increase the participation of the individual in his health. In this direction, nurse-led training and counseling programs are the leading methods that will increase the participation of patients in their health management, and research on this subject has been increasing in recent years. Jiang et al. In their study on patients with myocardial infarction, it was found that a nurse-led training and counseling program increased the quality of life and risk factor control. Boyne et al. In their study of heart failure patients, it was revealed that the knowledge, self-care, and self-efficacy of the patients increased after the intervention.

Despite growing evidence for the benefits of nurse-led education and counseling programs, no studies have been found with TAVI patients who might need this intervention the most. The aim of this study; is to examine the effect of education and follow-up program on quality of life, self-care, treatment compliance and hospital readmission in patients who underwent TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Transcatheter aortic valve implantation will be performed
* New York Health Association class II or III
* Mini-Mental Assessment test score ≥ 24
* Reachable by phone
* Volunteer to participate in the research
* Patients who can understand and speak Turkish

Exclusion Criteria:

* Stroke before and after the procedure
* Patients with kidney failure (to a level that requires dialysis treatment)
* Cancer (chemotherapy, radiotherapy)
* Chronic obstructive pulmonary disease (at a level that will require ventilation support)
* Severe hearing impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-18 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
EQ-5D (European QOL) Health Related Quality of Life Questionnaire | The scale will be applied on the first day of hospitalization, in the 1st and 3rd months to show the change in the patient's quality of life over the months.
  The EQ-5D scale was developed by the European Quality of Life (EuroQol) Working Group in 1990 for use in evaluative studies such as drug studies and policy research, and was revised in 1993. The EQ-5D defines health in terms of five sub-dimensions (mobility, self-care, general activities, pain/discomfort, and anxiety/depression) in a three-level structure as "no problem, moderately problematic, and severely problematic". An index score ranging from -0.59 to 1 is calculated from the 5 dimensions of the scale. In the score function, a value of 0 indicates death, a value of 1 indicates perfect health, while negative values indicate unconsciousness, being confined to a bed, etc. shows the situations.
European Heart Failure Self-Care Behaviors Scale | The scale will be applied on the first day of hospitalization, in the 1st and 3rd months to show the change in the patient's self care over the months.
  This scale was developed by Jaarsma et al. in 2003. The scale applied to measure the self-care behaviors of patients with heart failure has been determined as a scale that can be applied by the patients themselves, which does not require separate training and results in a short time. The scale consists of 12 items that include diagnosing symptoms related to heart failure such as edema, dyspnea, and self-care practices such as salt restriction or continuation of drug therapy. In the scoring of the scale, the participants are asked to choose one of the options for each item: I completely agree (1), agree (2), undecided (3), disagree (4), and completely disagree (5). The total score that can be obtained from the scale varies between 12-60. A high total score indicates low self-care, and a low score indicates high self-care.
Medication Adherence Report Scale | The scale will be applied on the first day of hospitalization, in the 1st and 3rd months to show the change in the patient's medication adherence over the months.
  The Medication Adherence Report Scale developed by Horne and Hankins (2001) to assess drug compliance, is a generic scale and can be customized according to the type of disease. Adaptations of the scale of many illnesses such as hypertension, diabetes, rheumatoid arthritis, asthma, chronic obstructive pulmonary disease, bipolar mood disorder, inflammatory bowel disease, hyperlipidemia and chronic pain are available in the literature. Participants are asked to indicate the frequency of occurrence of each of the five expressions. The scale is evaluated on a 5-point Likert-type scale with 5 = never, 4 = rarely, 3 = sometimes, 2 = often and 1 = very often. The total test score is obtained by summing the scores obtained from the items. Scores from the scale range from 5 to 25
Questionnaire | Hospitalization of TAVI patients due to cardiac causes within the first month after discharge will be considered as readmission.
  Hospital Readmission

CONTACTS AND LOCATIONS:
Overall Officials: Hatice MERT, Prof. Dr., Study Director — Dokuz Eylul University
Locations (1):
- Hospital of Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No